CLINICAL TRIAL: NCT03804528
Title: Assessing Cognitive Improvements, Brain Neuroplasticity and the Role of Genetic Factors After Aerobic Exercise in Sedentary Adults
Brief Title: Cognition and Neuroplasticity Sedentary Adults After 8 Weeks of Aerobic Exercise
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 Pandemic
Sponsor: University of Miami (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20180926; KL2TR002737 (NIH)
Record Dates: First submitted 2018-12-11; First posted 2019-01-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise group (All participants) (Experimental): Each participant will engage in 60 minute in-person daily sessions delivered 3 times/week for 8 consecutive weeks (a total of 24 sessions). Participants were provided with option to participate remotely due to COVID-19 pandemic.
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — Participants will be fitted with a heart rate monitor and will be instructed to walk (or trot) to maintain 55-64% of maximal heart rate (determined by exercise test) for the first 4-weeks of exercise or to maintain 65-90% of maximal heart rate (determined by exercise test) for the second 4-weeks of exercise during each session. Participants are provided the option to participate remotely due to COVID-19 pandemic, as detailed below. Both options are designed to be equivalent in intervention and outcome measures.
  Option A: Current, IRB-approved, in-person methods pending appropriateness based on current University of Miami recommendations and standard operating procedures as it relates to the COVID-19 pandemic.
  Option B: Remote option of current methods to maximize recruitment. This will be the only option until the study team obtains approval to resume Option A (as per University's safety guidelines).

SUMMARY:
The overall goal of the proposed study is to evaluate the effects of an 8-week aerobic exercise program on cognition and determine the relationship between cognitive improvements and Transcranial Magnetic Stimulation (TMS) neuroplasticity.

DETAILED DESCRIPTION:
The overall goal of the proposed study is to evaluate the effects of an 8-week aerobic exercise program on cognition and determine the relationship between cognitive improvements and neuroplasticity. The primary study aims include: 1) Quantify improvements in cognitive performance after 8 weeks (150 min per week) of moderate intensity aerobic exercise in sedentary adults ≥ 55 years of age; 2) Determine an association between changes in plasticity, aerobic capacity, and cognitive performance overall and by cognitive domain, after 8 weeks of moderate intensity aerobic exercise in sedentary adults ≥ 55 years of age.

Due to challenges posed by the COVID-19 pandemic, social distancing practices, and aiming to create a feasible scenario to continue the current study, we propose an additional option to safely adapt study methods to deliver the study in a home-based, fully remote manner. Importantly, this scenario also presents as an opportunity to collect meaningful data on our specific aims while translating this successful research program into a remote/home-based mode of delivery. A remote/home based option may also yield valuable preliminary data that will be relevant for planning future exercise studies in aging adults in the present "new normal". Therefore, this research project consist of two equivalent options:

Option A: Current, IRB-approved, in-person methods pending appropriateness based on current University of Miami recommendations and standard operating procedures as it relates to the COVID-19 pandemic.

Option B: Remote option of current methods to maximize recruitment. This will be the only option until the study team obtains approval to resume Option A (as per University's safety guidelines).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 55years
* no clinically detectable cognitive impairment (MoCA score ≥ 24 and Clinical Dementia Rating (CDR) score of 0)
* low activity level (individuals who do not engage in regular exercise, or currently exercise once a week or less)
* primary language is English

Exclusion Criteria:

* any unstable medical condition (i.e.: uncontrolled hypertension or uncontrolled diabetes)
* medical contraindication to physical exercise
* contraindication to TMS Neuroplasticity testing, as per the TMS Safety Guidelines.
* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG or family history of treatment resistant epilepsy
* Any current history of a psychiatric illness
* No medication is an absolute exclusion from TMS. Medications will be reviewed by the Principal Investigator and a decision about inclusion will be made based on the following:
* The subject's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination with other Central Nervous System (CNS) active drugs.
* The published TMS guidelines review medications to be considered with TMS.
* Any metal in the brain, skull or elsewhere unless approved by the responsible MD
* Any medical devices (i.e. Cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant, vagal nerve stimulator)
* Intracranial lesion
* Substance abuse or dependence within the past six months
* Pregnant women
* Vulnerable populations such as prisoner's
* People unable to consent themselves
* Subjects who, in the Investigator's opinion might not be suitable for the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce R Gomes-Osman, PT, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cabral DF, Hinchman CA, Nunez C, Rice J, Loewenstein DA, Cahalin LP, Rundek T, Pascual-Leone A, Gomes-Osman J. Harnessing Neuroplasticity to Promote Brain Health in Aging Adults: Protocol for the MOVE-Cog Intervention Study. JMIR Res Protoc. 2021 Nov 23;10(11):e33589. doi: 10.2196/33589. PMID 34817393

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise Group (All Participants): Each participant will engage in 60 minute in-person daily sessions delivered 3 times/week for 8 consecutive weeks (a total of 24 sessions).
  Aerobic Exercise in person: Participants will be fitted with a heart rate monitor and will be instructed to walk (or trot) to maintain 55-64% of maximal heart rate (determined by exercise test) for the first 4-weeks of exercise or to maintain 65-90% of maximal heart rate (determined by exercise test) for the second 4-weeks of exercise during each session.
  Option A: IRB-approved, in-person methods pending appropriateness based on current University of Miami recommendations and standard operating procedures as it relates to the COVID-19 pandemic.
  Option B: Remote option of current methods to maximize recruitment. This will be the only option until the study team obtains approval to resume Option A (as per University's safety guidelines).
Period: Overall Study
Arm/Group | Exercise Group (All Participants)
Started | 75
Completed | 52
Not Completed | 23
Not completed — Time Commitment | 18
Not completed — Health Reasons | 5

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics Data was collected and reported on those participants that completed the in-person and remote procedures.
Groups:
- Exercise Group (All Participants): Each participant will engage in 60 minute in-person daily sessions delivered 3 times/week for 8 consecutive weeks (a total of 24 sessions).
  Aerobic Exercise in person: Participants will be fitted with a heart rate monitor and will be instructed to walk (or trot) to maintain 55-64% of maximal heart rate (determined by exercise test) for the first 4-weeks of exercise or to maintain 65-90% of maximal heart rate (determined by exercise test) for the second 4-weeks of exercise during each session. Two equivalent options provided for participation, to accommodate for COVID-19 pandemic guidelines.
  Option A: Current, IRB-approved, in-person methods pending appropriateness based on current University of Miami recommendations and standard operating procedures as it relates to the COVID-19 pandemic.
  Option B: Remote option of current methods to maximize recruitment. This will be the only option until the study team obtains approval to resume Option A (as per University's safety guidelines).
Arm/Group | Exercise Group (All Participants)
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 7
  White | 24
  Hispanic | 17
  Hispanic/White | 3
  Asian | 1
BMI [Count of Participants; unit: Participants]
  Normal (18.5-24.9) | 14
  Overweight (25-29.9) | 19
  Obese Class I (30-34.9) | 13
  Obese Class 2 (35-39.9) | 6
Education Level [Count of Participants; unit: Participants]
  High School | 9
  Undergraduate/Associate Degree | 27
  Graduate Degree | 16
Health Status [Count of Participants; unit: Participants]
  Hospitalized | 41
  Taking prescribed medication | 41
  Smoking History | 13
  Alcohol Consumption | 41
  Caffeine consumption | 49
  Hypertension | 25
  Under beta-blocker | 6
  Arthritis or joint pain | 22
  Depression/anxiety | 13
  Thyroid disease | 12
  Lung/Asthma disease | 11
  Tumor or cancer | 10
  Migraine/Severe headache | 9
  Heart disease | 8
  Hearing loss | 6
  Fainting/Dizzy spells | 6
  Stomach/Intestinal disease | 4
  Diabetes | 4
MoCA - Montreal Cognitive Assessment Global Cognition [Mean (Standard Deviation); unit: units on a scale] — Montreal Cognitive Assessment or MoCA total scores. The Montreal Cognitive Assessment (MoCA) was initially developed as a test for mild cognitive impairment. It assesses seven areas of cognition for a maximal score of 30 (ranges 0-30). Higher scores indicate greater function.
  units on a scale | 26.4 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in TMS Plasticity Measures
Description: Index of the duration of the Theta-burst stimulation (TBS)-induced modulation of corticospinal excitability. This outcome measure refers to the identification of the time point (T5, T10, T15, T20 and T30). at which the normalized motor evoked potential (MEP) amplitude returns to baseline values (T0 or Baseline). This measure will be in Minutes Post Theta-Burst stimulation. This is a neurophysiological measure, and no group-based norms apply.
Time Frame: Baseline and Post-intervention (after 8 weeks of exercise)
Population: In 2020, due to challenges posed by the COVID-19 pandemic, social distancing practices, and aiming to create a feasible scenario to continue the study, an additional option was added to safely adapt study methods to deliver a home-based, fully remote program given that the duration of the pandemic was unknown at this time point. The study moved forward utilizing these two options, which were not designed as separate study arms but rather designed to be equivalent.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Exercise Group-All Participants: Each participant will engage in 60 minute in-person daily sessions delivered 3 times/week for 8 consecutive weeks (a total of 24 sessions).
  Aerobic Exercise in person: Participants will be fitted with a heart rate monitor and will be instructed to walk (or trot) to maintain 55-64% of maximal heart rate (determined by exercise test) for the first 4-weeks of exercise or to maintain 65-90% of maximal heart rate (determined by exercise test) for the second 4-weeks of exercise during each session.
  Option A: IRB-approved, in-person methods pending appropriateness based on current University of Miami recommendations and standard operating procedures as it relates to the COVID-19 pandemic.
  Option B: Remote option of current methods to maximize recruitment. This will be the only option until the study team obtains approval to resume Option A (as per University's safety guidelines).
Arm/Group | Exercise Group-All Participants
Number analyzed (Participants) | 29
minutes | 0.76 (0.47)

2. Primary Outcome: Cognitive Performance (RBANS)
Description: Cognitive performance will be assessed using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) a neuropsychological test battery in executive function, processing speed, learning, and language. It is made up of a series of twelve subtests that take approximately 30 minutes. For each of these, a lower number correct is indicative of a higher cognitive deficit. Subtests are their scales are: RBANS Semantic Fluency (0-unlimited), RBANS Picture Naming (0-10), RBANS List Learning (0-40), RBANS List Recall (0-10), RBANS Story Memory (0-24), RBANS Story Recall (0-12), RBANS List Recognition (0-20), RBANS Digit Span (0-16), RBANS Figure Recall (0-20), RBANS Coding (0-89), RBANS Figure Copy (0-20), RBANS Line Orientation (0-20).
Time Frame: Baseline and Post-intervention (after 8 weeks of exercise)
Population: Eligibility criteria met. Participants were considered at risk of cognitive decline due to their age, sedentary activity, and other lifestyle factors known to contribute to cognitive decline.
Measure: Mean (Standard Deviation); unit: mean total correct responses
Arm/Group | Exercise Group-All Participants
Number analyzed (Participants) | 52
mean total correct responses
  RBANS semantic fluency - Baseline | 20.6 (5.0)
  RBANS semantic fluency - Post-intervention | 20.3 (4.3)
  RBANS picture naming - Baseline | 9.4 (1.0)
  RBANS picture naming - Post-intervention | 9.6 (0.8)
  RBANS list learning - Baseline | 27.0 (4.7)
  RBANS list learning - Post-intervention | 28.7 (4.7)
  RBANS list recall - Baseline | 5.6 (2.3)
  RBANS list recall - Post-intervention | 6.4 (2.3)
  RBANS story memory - Baseline | 16.4 (3.6)
  RBANS story memory - Post-intervention | 17.3 (3.5)
  RBANS story recall - Baseline | 8.5 (2.5)
  RBANS story recall - Post-intervention | 8.9 (2.3)
  RBANS list recognition - Baseline | 18.6 (1.7)
  RBANS list recognition - Post-intervention | 19.2 (1.3)
  RBANS digital span - Baseline | 10.7 (2.2)
  RBANS digital span - Post-intervention | 10.8 (2.9)
  RBANS figure recall - Baseline | 14.1 (2.2)
  RBANS figure recall - Post-intervention | 14.1 (3.0)
  RBANS coding - Baseline | 43.8 (3.3)
  RBANS coding -Post-intervention | 44.0 (6.5)
  RBANS figure copy - Baseline | 15.8 (3.3)
  RBANS figure copy - Post-intervention | 16.3 (2.8)
  RBANS line orientation - Baseline | 17.4 (2.4)
  RBANS line orientation - Post-intervention | 17.2 (3.2)

3. Primary Outcome: Cognitive Performance (DKEFS)
Description: Cognitive performance will be assessed using a neuropsychological test battery in executive function, processing speed, learning, and language. The D-KEFS Verbal Fluency Test measures the ability to generate words fluently in an effortful phonemic format (letter fluency),from overlearned concepts (category fluency), and simultaneously shifting between overlearned concepts (category switching). Raw scores (correct responses, correct number of switches between categories) are converted to scaled scores with a mean of 10 and a standard deviation of 3. Higher scores reflect higher verbal fluency, and an increase in score pre-post would indicate improvement.
Time Frame: Baseline and Post-intervention (after 8 weeks of exercise)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Group (All Participants)
Number analyzed (Participants) | 52
score on a scale
  DKEFS letter fluency - Baseline | 10.9 (3.5)
  DKEFS letter fluency - Post-intervention | 11.4 (3.3)
  DKEFS category fluency - Baseline | 12.4 (2.9)
  DKEFS category fluency - Post-intervention | 11.5 (3.4)
  DKEFS category switching - Baseline | 12.5 (2.8)
  DKEFS category switching - Post-intervention | 12.7 (3.2)
  DKEFS category switching accuracy - Baseline | 12.7 (2.3)
  DKEFS category switching accuracy - Post-intervention | 12.8 (2.9)

4. Primary Outcome: Cognitive Performance (Digital Span)
Description: Digital span - Subtest of the Wechsler Adult Intelligence Scale fourth edition; Three sections: Digits Forward, Digits Backward, and Digits Sequencing. For each section, min. raw score value: 0; max. raw score value: 16. Higher the score, better the outcome.
Time Frame: Baseline and Post-intervention (after 8 weeks of exercise)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Exercise Group (All Participants)
Number analyzed (Participants) | 52
scores on a scale
  digital span forward - baseline | 10.2 (2.4)
  digital span forward - Post-intervention | 10.4 (2.3)
  digital span backward - baseline | 8.8 (2.2)
  digital span backward - post-intervention | 8.3 (2.4)
  digital span sequence - baseline | 8.7 (2.2)
  digital span sequence - post-intervention | 8.4 (2.3)

5. Secondary Outcome: Circulating Markers of Endothelium Function (BDNF)
Description: Blood samples will be collected to measure: brain-derived neurotrophic factor (BDNF) levels (measured as pg/mL).
Time Frame: Baseline
Population: COVID-19 PROVISIONS: Due to precautions required to prevent the spread of COVID-19, all in-person visits were discontinued; therefore, blood was not collected for all participants. Blood was only able to be collected for 24 participants at baseline.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Exercise Group-All Participants: Each participant will engage in 60 minute daily sessions delivered 3 times/week for 8 consecutive weeks (a total of 24 sessions).
  Aerobic Exercise: Participants will be fitted with a heart rate monitor and will be instructed to walk (or trot) to maintain 55-64% of maximal heart rate (determined by exercise test) for the first 4-weeks of exercise or to maintain 65-90% of maximal heart rate (determined by exercise test) for the second 4-weeks of exercise during each session.
Arm/Group | Exercise Group-All Participants
Number analyzed (Participants) | 24
pg/mL | 492.6 (348.1)

6. Secondary Outcome: Change in Cardiorespiratory Fitness
Description: Heart rate recovery (HRR) is the primary measure for cardiorespiratory fitness. HRR is defined as the change in the heart rate from the peak of exercise to the heart rate after 1-min (HRR-1) and 2-min test cessation (HRR-2).
Time Frame: Baseline and Post-intervention (after 8 weeks of exercise)
Population: Participants were considered at risk of cognitive decline due to their age, sedentary activity, and other lifestyle factors known to contribute to cognitive decline.
Measure: Mean (Standard Deviation); unit: heart beats per minute
Arm/Group | Exercise Group-All Participants
Number analyzed (Participants) | 52
heart beats per minute
  HRR1 - Baseline | 23.6 (11.6)
  HRR1 - Post-intervention | 27.0 (10.7)
  HRR2 - Baseline | 33.8 (12.5)
  HRR2 - Post-intervention | 40.4 (13.8)

7. Secondary Outcome: Circulating Markers of Endothelium Function (VEGF)
Description: Blood samples will be collected to measure vascular endothelial growth factor (VEGF) (measured as pg/mL).
Time Frame: Baseline
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Exercise Group (All Participants)
Number analyzed (Participants) | 24
pg/mL | 12.3 (5.4)

8. Secondary Outcome: Circulating Markers of Endothelium Function (Hs-CRP)
Description: Blood samples will be collected to measure high sensitivity C reactive protein (HS-CRP) (measured as mg/L).
Time Frame: Baseline
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Exercise Group (All Participants)
Number analyzed (Participants) | 24
mg/L | 1.9 (1.3)

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- Exercise Group (All Participants): Each participant will engage in 60 minute in-person daily sessions delivered 3 times/week for 8 consecutive weeks (a total of 24 sessions).
  Aerobic Exercise in person: Participants will be fitted with a heart rate monitor and will be instructed to walk (or trot) to maintain 55-64% of maximal heart rate (determined by exercise test) for the first 4-weeks of exercise or to maintain 65-90% of maximal heart rate (determined by exercise test) for the second 4-weeks of exercise during each session. Two equivalent options for in-person and remote participation were offered in response to the COVID-19 pandemic.
  Option A: Current, IRB-approved, in-person methods pending appropriateness based on current University of Miami recommendations and standard operating procedures as it relates to the COVID-19 pandemic.
  Option B: Remote option of current methods to maximize recruitment. This will be the only option until the study team obtains approval to resume Option A (as per University's safety guidelines, as mentioned above).
Arm/Group | Exercise Group (All Participants)
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic and resulting changes to remote clinical research modalities impacted the implementation of the study. Although the study was modified to accommodate remote participation, this modality prohibited the collection of clinical measures that required physical presence, such as TMS and blood collection, and required the adjustment for other measures, such as cardiorespiratory fitness assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT03804528/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT03804528/ICF_001.pdf